CLINICAL TRIAL: NCT04417114
Title: SystemIc iNflammation and Microvascular diSease PreventIon in psoRiatic diseasE
Acronym: INSPIRE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was not funded.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Marcelo F. Di Carli, MD, FACC, Chief Division of Nuclear Medicine and Molecular Imaging, Executive Director CV Imaging Program, Principal Investigator, Seltzer Family Professor of Radiology and Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BWH TBD
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis; Psoriatic Arthritis; Cardiovascular Risk Factor
Keywords: Coronary microvascular function
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single-Arm Open label (Experimental): This is a single-arm open label mechanistic clinical trial. Subjects will be treated with rosuvastatin at a dose of 20mg/day and uptitrated as tolerated to a dose of 40mg/day.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Statin
  Other Names: Crestor

SUMMARY:
This is a single-label open-arm mechanistic clinical study recruiting patients with psoriasis or psoriatic arthritis with elevated cardiovascular risk. Subjects enrolled in this study will receive statin treatment with rosuvastatin. The statin treatment in this study will be used as an intervention with widely known pleiotropic CV risk reduction effects, including anti-inflammatory reduction. Subjects will be studied before statin therapy and followed for 48 weeks on treatment. The primary outcome will be change in the coronary flow reserve (CFR) as measured by cardiac PET. Overall, this study will examine the impact of statin therapy on changes in CFR as a reflection of impaired coronary vasoreactivity and a manifestation of myocardial ischemia, which may precede clinical CV events (and visible changes in plaque morphology) in high-risk patients with psoriatic disease.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the impact of maximally tolerated statin (MTS) therapy on coronary flow reserve (CFR), reflecting coronary vasoreactivity and myocardial tissue perfusion. Impaired CFR is a manifestation of myocardial ischemia which may precede clinical CV events (and visible changes in plaque morphology) in high-risk patients with psoriatic disease. From previous studies, it is known that traditional risk factors underestimate cardiovascular risk in psoriatic disease. The central hypothesis of this study, is that MTS therapy - which has known pleiotropic CV risk reduction effects, including anti-inflammatory properties -- will quantitatively improve myocardial blood flow and CFR as measured by positron emission tomography (PET) over one year and reduce atherosclerotic burden, in patients with moderate-severe psoriasis or psoriatic arthritis. In so doing, improvement in coronary vasoreactivity, endothelial function, and tissue perfusion may have beneficial effects on myocardial mechanics, left ventricular deformation and function and, ultimately, symptoms and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years of age
* Documented evidence of PsO or PsA by a board-certified dermatologist or rheumatologist, respectively.
* Subjects on systemic therapy/phototherapy for PsO or PsA will be required to be on stable therapy for at least 3 months prior to enrollment

Plus, documented history of at least one of the following:

1. Hypertension
2. Obesity (BMI > 30)
3. Diabetes Mellitus
4. HsCRP > 3 mg/L within 30 days of enrollment

Exclusion Criteria:

* Patients on statin or PCSK9 inhibitor therapy, or use of statin therapy within the past year
* Documented history of other systemic inflammatory diseases, which in the opinion of the investigator would be inappropriate for enrollment.
* Prior history of untreated chronic infection (tuberculosis), severe fungal infection, or known HIV positive, chronic hepatitis B or C infection), prior history of solid malignancy, myeloproliferative or lymphoproliferative disease within 5 years, excluding treated non-melanoma skin cancer
* NYHA class IV heart failure
* Active liver disease including unexplained, persistent elevations of serum transaminases or serum transaminase elevation > 3 x the upper limit of normal.
* Severe renal impairment
* Pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Coronary Flow Reserve (CFR) | Baseline and 12 months
  CFR will be measured by cardiac PET at baseline prior to initiating treatment and following 12 months of statin therapy.

SECONDARY OUTCOMES:
Change in the total coronary plaque burden measured by cardiac CT angiography (CCTA) | Baseline and 12 months
  Total coronary plaque burden will be assess by CCTA at baseline and following 12 months of statin therapy
Change in change in LV peak global longitudinal strain (GLS) (systolic function), measured by transthoracic echocardiogram (TTE) | Baseline and 12 months
  GLS will be measured by TTE at baseline and following 12 months of statin therapy
Change in tissue Doppler mitral annular early diastolic relaxation velocity (E') (diastolic function), measured by transthoracic echocardiogram (TTE) | Baseline and 12 months
  E' will be measured by TTE at baseline and following 12 months of statin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Di Carli, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No